CLINICAL TRIAL: NCT02315495
Title: Combining Saxagliptin and Acarbose to Improve Postprandial Glycaemia in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zilin Sun (Other)
Responsible Party: Sponsor-Investigator, Zilin Sun, MD, PhD of Department of Endocrinology, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ISSSAXA0015
Record Dates: First submitted 2014-12-03; First posted 2014-12-12 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 5 mg saxagliptin + 100 mg acarbose (Experimental): Acute dosing:
  5 mg saxagliptin is given with water, 60 min before a test meal 100 mg acarbose is given with a test meal
  Interventions: Drug: Saxagliptin; Drug: Acarbose
- 5 mg saxagliptin (Experimental): Acute dosing:
  5 mg saxagliptin is given 60 min before a test meal,
  Interventions: Drug: Saxagliptin
- 100 mg acarbose (Experimental): Acute dosing:
  100 mg acarbose is given with a test meal
  Interventions: Drug: Acarbose
- control (No Intervention)

INTERVENTIONS:
Drug: Saxagliptin
  Other Names: Onglyza
  Arms: 5 mg saxagliptin; 5 mg saxagliptin + 100 mg acarbose
Drug: Acarbose
  Other Names: Glucobay
  Arms: 100 mg acarbose; 5 mg saxagliptin + 100 mg acarbose

SUMMARY:
The proposed study is designed to evaluate (i) the effects of saxagliptin, with or without acarbose, on gastric emptying, postprandial glycaemia, and plasma intact GLP-1, insulin, C-peptide and glucagon after a high carbohydrate meal, and (ii) whether the magnitude of the effects of saxagliptin and/or acarbose is related to the rate of gastric emptying, in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (World Health Organisation (WHO) criteria), managed by diet alone (i.e. no oral hypoglycaemic drugs or insulin)
* Body mass index (BMI) 20 - 40 kg/m2
* Age 18 - 70 years
* Males and post-menopausal females (to control for the effect of the menstrual cycle on gut hormone secretion)
* Glycated haemoglobin A1c (HbA1c) ≥ 6.0% and ≤ 7.9%
* Haemoglobin above the lower limit of the normal range (i.e. >135g/L for men and 115g/L for women), and ferritin above the lower limit of normal (i.e. >10mcg/L)

Exclusion Criteria:

* Use of any medication that may influence gastrointestinal motor function, body weight or appetite
* Evidence of drug abuse, consumption of more than 20 g alcohol or 10 cigarettes on a daily basis
* History of gastrointestinal disease, including significant upper or lower gastrointestinal symptoms, pancreatitis, or previous gastrointestinal surgery (other than uncomplicated appendicectomy or cholecystectomy)
* Other significant illness, including epilepsy, cardiovascular or respiratory disease
* Autonomic nerve damage (as assessed by standardised cardiovascular reflex tests [36])
* Impaired renal or liver function (as assessed by calculated creatinine clearance < 90 mL/min or abnormal liver function tests (> 2 times upper limit of normal range))
* Allergy to vildagliptin or any other 'gliptin'
* Donation of blood within the previous 3 months
* Participation in any other research studies within the previous 3 months
* Females who are pre-menopausal
* Inability to give informed consent
* Vegetarians

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-04-03; Primary Completion 2016-08-26 (Actual); Study Completion 2016-08-26 (Actual)

PRIMARY OUTCOMES:
Blood glucose concentrations at pre-defined intervals | -60,-10,0,30,60,90,120,180min

SECONDARY OUTCOMES:
Plasma concentrations of incretin hormones at pre-defined intervals | -60,-10,0,30,60,90,120,180min
Plasma concentrations of insulin at pre-defined intervals | -60,-10,0,30,60,90,120,180min
Plasma concentrations of C-peptide at pre-defined intervals | -60,-10,0,30,60,90,120,180min
Plasma concentrations of glucagon at pre-defined intervals | -60,-10,0,30,60,90,120,180min
half-emptying time (T50) | 0-180min

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Zhongda Hospital. Institute of Diabetes, Southeast University, Nanjing, Jiangsu, China